CLINICAL TRIAL: NCT00920361
Title: Designated Drug Use Investigation 1 of Follistim Injection
Brief Title: Designated Drug Use Investigation 1 of Follistim Injection (Study P06130)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06130
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Fertilization in Vitro
MeSH Terms: interventions — follitropin beta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who underwent IVF
  Interventions: Drug: Follitropin beta

INTERVENTIONS:
Drug: Follitropin beta — Normally, Follistim Injection 150 or 225 IU will be administered (s.c. or i.m.) once a day for 4 days as follitropin beta (genetical recombination). The dosage will be adapted to growth of follicles (75-375 IU for 6-12 days, in general). If more than 3 follicles of mean diameter 16-20 mm are confirmed by ultrasound tomography, ovulation will be stimulated by using Human Chorionic Gonadotropin (hCG) drugs.

SUMMARY:
To evaluate dosage and administration method, efficacy and safety of Puregon and the relationship between background factors of patients and dose and administration method.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent IVF

Exclusion Criteria:

* Patients with tumors of ovary, breast, uterus, pituitary or hypothalamus
* Pregnant or possible pregnant women, or lactating women
* Patients with undiagnosed atypical vaginal bleeding
* Patients with a history of hypersensitivity to any of the ingredients of this product.
* Patients with ovarian cysts or enlarged ovaries, not related to polycystic ovarian disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese 1100 patients
Sampling Method: Non-Probability Sample
Enrollment: 1664 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 2 months, from initiation of treatment to confirmation of pregnancy.

SECONDARY OUTCOMES:
Pregnancy outcome | 2 months, from initiation of treatment to confirmation of pregnancy.